CLINICAL TRIAL: NCT05338541
Title: Tucidinostat Plus Etoposide in the Treatment of Relapsed or Refractory Neuroblastoma in Children
Brief Title: Tucidinostat Plus Etoposide in the Treatment of Neuroblastoma in Childhood.
Acronym: CSIIT-Q36
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yizhuo Zhang (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Zhang, Director of department of pediatric cancer,Principal Investigator,Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIDA-01
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Neuroblastoma in Children
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucidinostat and etoposide (Experimental)
  Interventions: Drug: Tucidinostat and etoposide

INTERVENTIONS:
Drug: Tucidinostat and etoposide — Tucidinostat: 3+3 design，14 mg/m2，17.5 mg/m2，23 mg/m2 etoposide: 50mg/m2,

SUMMARY:
Neuroblastoma is a malignant tumor that develops in infants and kids. Dysregulation of histone acetylation is associated with a series of malignant tumors. Neuroblastoma is caused by defective neural crest differentiation due to abnormal gene regulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3~18 years old;
2. Patients must have a life expectancy of at least 6 weeks and a Lansky (≤16 years) or Karnofsky (>16 years) score of at least 50;
3. Histologically confirmed neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines;
4. Patients must have a history of high-risk neuroblastoma, at least one measurable lesions according to the RECIST 1.1;
5. Patients who have progressed, recurrent or refractory disease after first-line treatment;
6. The residual disease biopsy must be done, if patiens who have persistent disease obtain incomplete response after first line treatment;
7. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study registration；
8. Patients have not received enzyme-induced anticonvulsant therapy;
9. Patients have not received valproic acid within 30 days before admission;
10. ANC ≥ 1.5×10^9/L, PLT ≥75×10^9/L;TBIL≤1.5ULN, ALT and AST≤3×ULN（ALT and AST≤5×ULN if liver metastasis）;BUN and Cr≤1.5×ULN 9）LVEF ≥ 50% and QTc≤470 ms.
11. Patients' guardians must be willing and able to understand and comply with the protocol for the duration of the study.

Exclusion Criteria:

1. Patients with severe cardiovascular disease;
2. Patients who have previously received organ transplants;
3. Inability to swallow pills;
4. Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
5. Active HIV, hepatitis B or hepatitis C;
6. Researchers believe that patients are unsuitable for any other situation in this study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 1 year
  Dose-limiting toxicity defined as any Grade 4 hematological toxicity and any > Grade 3 non-hematologic toxicity.
Maximum Tolerated Dose (MTD) | 1 year
  Maximum tolerated dose is highest dose level in which 6 patients treated with at most 1 experiencing DLT.

SECONDARY OUTCOMES:
Response Rate(ORR) | 2 years
  Objective Response Rate（ORR）by RECIST 1.1,the total proportion of patients with complete response（CR）, partial response（PR）
progression-free survival (PFS) | 2 years
  Time from treatment until disease progression or death
overall survival (OS) | 2 years
  Time from treatment until death from any cause
disease control rate (DCR) | 2 years
  The total proportion of patients with complete response（CR）, partial response（PR）and Stable Disease（SD）

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Yizhuo, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No